CLINICAL TRIAL: NCT01200706
Title: Clinical Efficacy of Amoxicillin Given Twice or Three Times a Day Among Children With Non-severe Community-acquired Pneumonia
Brief Title: Clinical Efficacy of Amoxicillin Given Twice or Three Times a Day Among Children With Non-severe Pneumonia
Acronym: PNEUMOPACEf
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federal University of Bahia (Other)
Responsible Party: Prof. Cristiana Maria Costa Nascimento-Carvalho, Federal University of Bahia School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APR0127/2006
Record Dates: First submitted 2010-09-13; First posted 2010-09-14 (Estimated); Last update posted 2011-07-20 (Estimated); Status verified 2010-09

CONDITIONS: Community-acquired Pneumonia
Keywords: children aged under 5 years; Non-severe
MeSH Terms: conditions — Community-Acquired Pneumonia | interventions — Amoxicillin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Amoxicillin given twice a day (Active Comparator)
  Interventions: Drug: Amoxicillin
- Amoxicillin given three times a day (Active Comparator)
  Interventions: Drug: Amoxicillin

INTERVENTIONS:
Drug: Amoxicillin — amoxicillin 50mg/kg/day given in two different administration schemes
  Other Names: Placebo with amoxicillin,in the opposite posologic scheme

SUMMARY:
The purpose of the study is to compare the clinical efficacy of amoxicillin given twice or three times a day to children with non-severe community-acquired pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 2 and 59 months
* Report of respiratory complaints
* Presence of pulmonary infiltrate on chest x-ray taken on admission and read by the pediatrician on duty

Exclusion Criteria:

* lower chest indrawing
* danger signs (inability to drink, convulsions, somnolence, central cyanosis, grunting in a calm child)
* diagnosed underlying chronic diseases (anatomic abnormalities of the respiratory tract, chronic pulmonary illness besides asthma, immunological defects, progressing neurological disorders, psychomotor retardation, heart disease with clinical repercussion, hemoglobinopathy, liver or kidney disease)
* severe malnutrition
* other concurrent infection
* hospitalization during the previous 7 days
* amoxicillin or similar antibiotic use during the last 48 hours
* allergy to amoxicillin
* history of aspiration

Ages: 2 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 820 (Actual)
Dates: Start 2006-11; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
clinical efficacy | 48 hours
  resolution of fever, difficulty breathing and tachypnea

SECONDARY OUTCOMES:
Resolution of cough | 96 hours
  Disappearance of cough

CONTACTS AND LOCATIONS:
Overall Officials: Cristiana M Nascimento-Carvalho, MD, PhD, Principal Investigator — Federal University of Bahia School of Medicine
Locations (1):
- Professor Hosannah de Oliveira Pediatric Center, Salvador, Estado de Bahia, Brazil

REFERENCES:
- [Derived] Nascimento-Carvalho AC, Vilas-Boas AL, Fontoura MH, Vuorinen T, Nascimento-Carvalho CM; PNEUMOPAC-Efficacy Study Group. Respiratory viruses among children with non-severe community-acquired pneumonia: A prospective cohort study. J Clin Virol. 2018 Aug;105:77-83. doi: 10.1016/j.jcv.2018.06.003. Epub 2018 Jun 6. PMID 29908521
- [Derived] Nascimento-Carvalho AC, Vilas-Boas AL, Fontoura MH, Xu M, Vuorinen T, Soderlund-Venermo M, Ruuskanen O, Nascimento-Carvalho CM; PNEUMOPAC-Efficacy Study Group. Serologically diagnosed acute human bocavirus 1 infection in childhood community-acquired pneumonia. Pediatr Pulmonol. 2018 Jan;53(1):88-94. doi: 10.1002/ppul.23891. Epub 2017 Oct 13. PMID 29028159
- [Derived] Nascimento-Carvalho CM, Xavier-Souza G, Vilas-Boas AL, Fontoura MH, Barral A, Puolakkainen M, Ruuskanen O; PNEUMOPAC-Efficacy Study Group. Evolution of acute infection with atypical bacteria in a prospective cohort of children with community-acquired pneumonia receiving amoxicillin. J Antimicrob Chemother. 2017 Aug 1;72(8):2378-2384. doi: 10.1093/jac/dkx126. PMID 28475737
- [Derived] Vilas-Boas AL, Fontoura MS, Xavier-Souza G, Araujo-Neto CA, Andrade SC, Brim RV, Noblat L, Barral A, Cardoso MR, Nascimento-Carvalho CM; PNEUMOPAC-Efficacy Study Group. Comparison of oral amoxicillin given thrice or twice daily to children between 2 and 59 months old with non-severe pneumonia: a randomized controlled trial. J Antimicrob Chemother. 2014 Jul;69(7):1954-9. doi: 10.1093/jac/dku070. Epub 2014 Mar 19. PMID 24648506
- [Derived] Xavier-Souza G, Vilas-Boas AL, Fontoura MS, Araujo-Neto CA, Andrade SC, Cardoso MR, Nascimento-Carvalho CM; PNEUMOPAC-Efficacy Study Group. The inter-observer variation of chest radiograph reading in acute lower respiratory tract infection among children. Pediatr Pulmonol. 2013 May;48(5):464-9. doi: 10.1002/ppul.22644. Epub 2012 Aug 8. PMID 22888091